CLINICAL TRIAL: NCT02734849
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Study to Evaluate Multiple Doses of AK001 in Patients With Moderate to Severe Nasal Polyposis
Brief Title: Study to Evaluate Multiple Doses in Patients With Nasal Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK001-002
Record Dates: First submitted 2016-03-24; First posted 2016-04-12 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2018-12

CONDITIONS: Nasal Polyposis
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 mg AK001 (Experimental): 25 mg AK001 will be administered as multiple doses
  Interventions: Drug: AK001 low dose
- 250 mg AK001 (Experimental): 250 mg AK001 will be administered as multiple doses
  Interventions: Drug: AK001 high dose
- Placebo (Placebo Comparator): A placebo comparator consisting of inactive excipients will be administered as multiple doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK001 low dose — 25 mg AK001 will be administered as multiple doses
  Arms: 25 mg AK001
Drug: AK001 high dose — 250 mg AK001 will be administered as multiple doses
  Arms: 250 mg AK001
Drug: Placebo — Placebo will be administered as multiple doses
  Arms: Placebo

SUMMARY:
This is a phase 2 study to evaluate multiple doses of AK001 across 2 active doses. Pharmacodynamic activity will also be evaluated.

DETAILED DESCRIPTION:
AK001 is a monoclonal antibody which may be useful in the treatment of patients with moderate to severe nasal polyposis

ELIGIBILITY:
Inclusion Criteria:

* TPS of ≥5 for both nostrils with presence on endoscopy of nasal polyps of grade ≥2 in each nostril according to the polyp grading scale
* History of sinusitis symptoms
* SNOT-22 ≥30
* No clinically significant Screening 12-lead ECG, vital sign, hematology, chemistry, or urinalysis findings

Exclusion Criteria:

* Use of systemic corticosteroids within 6 weeks of screening
* Chronic use of antibiotic therapy within 3 months prior to Screening
* Nasal surgery (including polypectomy) within 6 months prior to Screening
* Use of investigational drugs or participation in another clinical trial within 30 days prior to Screening or 5 half-lives, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, Principal Investigator — University Hospital, Ghent
Locations (15):
- United States (5):
  - Investigator site, Chicago, Illinois
  - Investigator site, Boston, Massachusetts
  - Investigator site, Pittsburgh, Pennsylvania
  - Investigator site, Houston, Texas
  - Investigator site, Charlottesville, Virginia
- Belgium (2):
  - Investigator site, Ghent
  - Investigator site, Leuven
- Germany (2):
  - Investigator site, Düsseldorf
  - Investigator site, Münster
- Investigator site, Amsterdam, Netherlands
- Spain (3):
  - Investigator site, Barcelona
  - Investigator site, Jerez de la Frontera
  - Investigator, Valencia
- United Kingdom (2):
  - Investigator site, Cambridge
  - Investigator site, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date First Patient First Visit 04 April 2016 Date Last Patient Last Visit 05 January 2018 Date Enrollment was Terminated 31 May 2017
Groups:
- 25 mg AK001: 25 mg AK001 was administered as a single IV infusion through a peripheral vein on Days 0, 21, and 49.
- 250 mg AK001: 250 mg AK001 was administered as a single IV infusion through a peripheral vein on Days 0, 21, and 49.
- Placebo: Placebo was administered as a single IV infusion through a peripheral vein on Days 0, 21, and 49.
Period: Overall Study
Arm/Group | 25 mg AK001 | 250 mg AK001 | Placebo
Started | 16 (One patient was randomized but never received study treatment and excluded from all analysis sets.) | 14 | 10
Completed | 12 | 14 | 9
Not Completed | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg AK001 | 250 mg AK001 | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 10 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 10 | 37
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Median (Full Range); unit: Years] | 48.0 [24 to 71] | 46.5 [27 to 63] | 45.0 [29 to 60] | 45.0 [24 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 18
  Male | 10 | 6 | 5 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 14 | 10 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 14
  Europe | 10 | 9 | 6 | 25
Total Polyp Score (TPS) [Median (Full Range); unit: units on a scale] | 6.0 [4 to 8] | 6.0 [4 to 8] | 6.0 [4 to 8] | 6.0 [4 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Polys Score (TPS)
Description: NPS was the sum of the right and left nostril scores, as evaluated by means of nasal endoscopy. Change in TPS from Baseline (prior to the first dose) to Week 12 (Day 84) was the primary outcome of the study. TPS ranges from 0 to 8 (scored 0 [no polyp] to 4 [large polyps] for each nostril), with a lower score indicating smaller-sized polyps, a higher scores mean a worse outcome.
Time Frame: From Baseline (prior to the first dose) to Week 12 (Day 84)
Population: Modified Intent-to-Treat (MITT) population included all randomized subjects who have taken at least one dose of the study drug and had both a baseline and at least one post-baseline efficacy assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 25 mg AK001 | 250 mg AK001 | Placebo
Number analyzed (Participants) | 15 | 14 | 10
score on a scale | -0.5 [-1.3 to 0.3] | -0.3 [-1.1 to 0.5] | -0.2 [-1.1 to 0.7]

ADVERSE EVENTS:
Time Frame: The time of study drug administration until completion of the last study-related procedure at approximately 24 weeks, i.e. Day 168, or early termination of the study.
Description: If a patient completed the study with an ongoing adverse event (AE), investigational site personnel continued to follow-up until AE resolution and the documentation thereof. If, after 30 days from the study completion date, the AE was still continuing but not assessed as serious, the outcome was recorded as ongoing.
Arm/Group | 25 mg AK001 | 250 mg AK001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 11/15 | 10/14 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg AK001 (N=15) | 250 mg AK001 (N=14) | Placebo (N=10)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (3) | 1 (2)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
After 40 of the 70 patients planned were randomized in the study, enrollment was stopped as the Sponsor decided not to pursue further development of AK001. The study was not stopped for any safety concern. Early termination resulted uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT02734849/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02734849/SAP_001.pdf